CLINICAL TRIAL: NCT04818879
Title: Electromyographic Response Control in the Application of Vojta Therapy in the Abdominal Muscles of Healthy Young Adults
Brief Title: Abdominal Electromyographic Control in Vojta Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Collaborators: Colegio Profesional de Fisioterapeutas de Castilla y León (Unknown)
Responsible Party: Principal Investigator, Pérez-Robledo, Fátima, Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NEUROUSAL04/2021
Record Dates: First submitted 2021-03-21; First posted 2021-03-26 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Abdominal Muscles
Keywords: Electromyography; Abdominal Muscles; Muscle Contraction; Outcome and Process Assessment; Health Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental)
  Interventions: Other: Vojta
- Control group (Sham Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Vojta — The subject will be placed on a stretcher with the torso uncovered. Once the adhesive electrodes have been placed in the different recording areas on the anterior part of the trunk, a recording of the activity at rest will begin, two minutes of stimulation (digital pressure), one minute of rest, two minutes of stimulation in the contralateral side and, finally, one minute of rest.
  The therapy consists of the application of a stimulating pressure in the pectoral area in the pattern of the locomotion complex of reflex rolling in its first phase. For this, the subject will be placed in a supine position aligned with respect to the axial axis, with the arms along the body, the lower extremities in extension, and the head extended with a rotation of approximately 30º towards one side of the stimulation. The manual stimulation pressure will be exerted in the space between the 6th-7th or the 7th-8th rib under the mammillary line, with a force of about 2 kg.
  Arms: Interventional group
Other: Control — The subject will be placed on a stretcher with the torso uncovered. Once the adhesive electrodes have been placed in the different recording areas on the anterior part of the trunk, a recording of the activity at rest will begin, two minutes of stimulation (digital pressure), one minute of rest, two minutes of stimulation in the contralateral side and, finally, one minute of rest.
  The control group will receive an application in an area with low receptor density located on the thigh, with a force of about 2 kg.
  Arms: Control group

SUMMARY:
A randomized clinical trial on a cohort of healthy subjects of legal age, both sexes, recruited from the university community and who will be randomly distributed into two groups (experimental and control). The objective will be to determine the feasibility of the standardized intervention protocol on the stabilizing muscles of the trunk (external oblique and internal oblique) before, during and after the application of Vojta Therapy, and to know the effects produced on the Musculature studied after performing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Full cognitive capacity.

Exclusion Criteria:

* Subjects with neuro-muscular pathologies that affect the abdominal muscles, previous surgeries in the area or any chronic neurological or organic disorder that may alter the results.
* Vaccinated in the 10 days prior to the intervention
* Fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Electromyographic activity in abdominal muscles | Change from Baseline electromyographic activity at 7 minutes.
  The electromyographic activity of internal and external obliques in nanovolts will be collected before, during and after the intervention.

SECONDARY OUTCOMES:
Date of birth | Baseline
  It will be registered at the beginning of the study in order to calculate the age of the participant.
Sex | Baseline
  It will be registered at the beginning of the study.
Height | Baseline
  It will be registered at the beginning of the study in centimeters.
Weight | Baseline
  It will be registered at the beginning of the study in kilograms.
International Physical Activity Questionnaire | Baseline
  It will be measured at the beginning of the study to quantify the level of physical activity of the participant. This validated scale allows you to determine if you have a low, moderate or high physical level.

CONTACTS AND LOCATIONS:
Overall Officials: Fátima Pérez-Robledo, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided